CLINICAL TRIAL: NCT07219940
Title: An Open-label and Dose-escalation Phase I Clinical Study to Evaluate the Tolerability, Safety, and Pharmacokinetics of HLA-G-targeted Exosome (SOB100) in Healthy Subjects
Brief Title: A Study to Investigate HLA-G Targeted Exosome (SOB100) in Healthy Subjects
Acronym: αHLA-G Exo-01
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shine-On Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOB100-CL-Proto-01
Record Dates: First submitted 2025-10-19; First posted 2025-10-22 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-10

CONDITIONS: Healthy Subjects; Exosome; Targeted Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SOB100 (Experimental)
  Interventions: Drug: SOB100

INTERVENTIONS:
Drug: SOB100 — Drug: SOB100 Participants will receive SOB100 and evaluate the safety and tolerability of SOB100 during the dose escalation phase.

SUMMARY:
The investigational drug, SOB100, is an HLA-G targeted exosome equipped with a nanobody namely anti-HLA-G VHH on the exosome membrane. This is a Phase I dose escalation study to exam the tolerability, safety, and pharmacokinetics in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥ 18 years old
2. Overtly healthy subject, who is considered to be generally healthy based on medical history, 12-lead ECG, and physical examinations, as judged by the Investigator
3. Able to understand and comply with procedures in the protocol as judged by Investigator and sign the informed consent form (ICF)
4. Adequate organ function

Exclusion Criteria:

1. With known or suspected to be hypersensitivity to HLA-G related treatment.
2. Confirmed active HIV, HBV, or HCV infection
3. With active fungal, bacterial, viral or atypical infection requiring systemic medication
4. History of cancer (malignancy) or have ever received any anti-cancer therapy
5. Has ever received cell therapy or organ transplantation
6. Substance abuse or addictive use of drugs for nonmedical purposes
7. Female subject is lactating, has a positive pregnancy test or refuse to practice highly effective contraception
8. Male subjects with a female spouse/partner who is of childbearing potential refuse to adopt at least one highly effective method of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse event (AE) | From start until 3 weeks after the last dose of SOB100
Incidence of serious adverse event (SAE) | From start until 3 weeks after the last dose of SOB100
Incidence of treatment-emergent adverse event (TEAE) | From start until 3 weeks after the last dose of SOB100
Abnormalities in physical examination (PE) | From start until 3 weeks after the last dose of SOB100
Abnormalities in ECG | From start until 3 weeks after the last dose of SOB100

OTHER OUTCOMES:
Area Under the Curve of SOB100 (AUC) | From baseline to 3 weeks after the last dose of SOB100
  Pharmacokinetics (PK) parameters
Maximum observed plasma concentration of SOB100 (Cmax) | From baseline to 3 weeks after the last dose of SOB100
  Pharmacokinetics (PK) parameters
Half-life of SOB100 (T1/2) | From baseline to 3 weeks after the last dose of SOB100
  Pharmacokinetics (PK) parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Parexel International - Baltimore Early Phase Clinical Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No